

#### **Letter of Information**

## The Effect of Different Time-restricted Eating Windows on Body Composition

Bryce Knapp- Undergraduate researcher 807-620-0441 Peter Lemon- Exercise Nutrition Research Laboratory Principal investigator 661-2111, ext 88139

You are being invited to participate in this study because you responded to our advertisement. This letter provides you with detailed information about our study which will be conducted in the Exercise Nutrition Research Laboratory (Rm 2235 3M Centre) so you can decide if you would like to participate. The data obtained will be used to complete requirements for Kinesiology 4443 – an undergraduate research course.

#### Introduction

Having a higher percentage of body fat has several significant adverse health effects which diminish with fat loss. Eating patterns have changed over human evolution and there is some evidence that an intermittent pattern of eating, i.e., one with periods of fasting interspersed similar to how our distant ancestors likely ate, is better for both losing fat and maintaining healthy body fat stores than a more regular eating pattern (3 or more meals a day). This research study is designed to provide information of whether the time of the eating period effects body composition. Please read this letter carefully and ask any questions that you have before agreeing to participate in this study.

## **Purpose**

To determine if the timing of an 8-hour eating window will affect body composition.

#### **Description**

This study requires you to do the following:

- Restrict your eating to an 8-hour time period (eat whatever you like between 6am-2pm or 2pm- 10pm at least 5 days a week)
- Drink only zero calorie beverages (coffee, tea, water) outside the feeding window.
- Have participants answer a questionnaire and check a box for which days during the week the participant complied with the protocol.
- Have your body composition (fat and lean body mass) measured using non-invasive densitometry (Bod Pod this requires you to sit in a chamber while the space [volume] your body takes up is assessed). This along with your body mass allows us to calculate your body density and your body composition one week prior to and after 4 weeks of time restricted eating. The procedure takes about 5 minutes.



#### **Benefits**

Participation in this study may not be of any direct benefit to you, although you might lose body fat which is associated with many positive health benefits and you will find out how these types of research studies are conducted. Further, the results of this study may provide important information that will help fight against the rising incidence of obesity which has become a significant health problem in all developed countries.

## **Risks**

This study has minimal risks. First, you may feel minor hunger sensations for the first few days. Further, in rare cases you could experience headaches, sleep disruption, heartburn, weakness, lack of focus and/or concentration during the first few days as your body adjusts to the new eating pattern. All of these are considered minor with no lasting effects.

## You can participate in this study if you:

- are 18-25 years of age

## You CANNOT participate in this study if you:

- have symptoms or take medication for respiratory, cardiovascular, neuromuscular, or metabolic disease (self-reported)
- Are pregnant or become pregnant (self-reported)
- Have a body mass index less than 26
- No personal history of intermittent fasting in the past 6 months (self-reported)
- No diabetes (self-reported)

#### Time Involved

If you choose to take part in this study, your time commitment will be minimal as follows:

- you will report to room 2235 3M Centre on main campus for an initial 10-minute orientation session discussing consent and study information.
- you will report for 4 body composition evaluation periods (approximately 15 minutes each)
- Fill out two biweekly questionaries' regarding adherence to the protocol.

## **Voluntary Participation**

Participation in this study is voluntary. You may refuse to participate, refuse to answer any questions, or withdraw from the study at any time with no effect on your academic or employment status. Should you become pregnant you will be excused from the study. Further, the investigators have the right to withdraw you from the study at any time for reasons related to you (e.g., not following the study-related directions) or because the entire study has been stopped. Data from participants that choose to withdraw from the study will be removed from the database system while maintaining participant confidentiality.

## **Confidentiality**

Although your name and email addresses will be collected to allow for scheduling of testing sessions, these data will not be stored at the conclusion of the study, unless you

agree to being contacted for future studies after this study is completed. When the results of this study are reported, they will be coded to protect your identity and privacy. Individual results will be held in strict confidence and all data will be stored behind a firewall and will be encrypted. Only the investigators will have access to your records. Your data will be kept indefinitely for comparison with future studies but de-identified so no one will be able to link the results to you. You are encouraged to ask questions of the investigators regarding the purpose of the study or any of the methods to be used.

Representatives of the University of Western Research Ethics Board may contact you or require access to your study-related records to monitor conduct of the research.

## **Inquiries Concerning the Study**

If you have any questions about this study or your care/treatment please contact:

Bryce Knapp- Undergraduate investigator (<u>bknapp3@uwo.ca</u>)
Peter Lemon – Principal investigator (<u>plemon@uwo.ca</u>)

If you have questions about the conduct of this study or your rights as a research participant you may contact: 519-661-3059 or by email at <a href="mailto:ethics@uwo.ca">ethics@uwo.ca</a> Office of Research Ethics, Western University.

You will be given a copy of this letter of information and consent form once it has been signed. You do not waive any legal rights by signing the consent form.

## CONSENT FORM

# The Effect of Different Time-restricted Eating Windows on Body Composition

| I, | ture of the study explain | |
|---|---|---|
| Please indicate if you would like to be in the appropriate box below: | n to be retained for contac | t about future studies. |
| Participant's Name:(Print name he | ere) | (Signature) |
| Date: | | |
| Person Obtaining Informed Consent: | (Print Name here) | (Signature) |
| Date: | | |